CLINICAL TRIAL: NCT07377734
Title: A Multicenter, Randomized, Open-Label, Controlled Clinical Trial of Intrauterine Injection of Recombinant Humanized Type III Collage in the Fertility-Sparing Treatment of Endometrial Cancer or Atypical Hyperplasia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wang Jianliu (Other)
Responsible Party: Sponsor-Investigator, Wang Jianliu, Professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHD014-001
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Atypical Endometrial Hyperplasia; Endometrial Cancer
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Progestins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this arm will receive a combination therapy of oral high-dose progestin and intrauterine injections of Recombinant Humanized Type III Collagen Lyophilized Fibers for fertility preservation
  Interventions: Drug: Recombinant Humanized Type III Collagen Lyophilized Fibers + High-dose Progestin
- Control Group (Active Comparator): Participants in this arm receive the current standard-of-care treatment for fertility preservation in endometrial cancer, which consists of oral high-dose progestin alone. This allows for a direct comparison of efficacy and safety between the progestin-only therapy and the progestin-collagen combination therapy
  Interventions: Drug: High-dose Progestin

INTERVENTIONS:
Drug: Recombinant Humanized Type III Collagen Lyophilized Fibers + High-dose Progestin — Participants in this group will receive a combination therapy. They will take oral high-dose progestin (Medroxyprogesterone Acetate 250mg-500mg/d or Megestrol Acetate 160mg-320mg/d) daily. Additionally, they will receive three intrauterine submucosal injections of Recombinant Humanized Type III Collagen Lyophilized Fibers (50mg per injection) via hysteroscopy at months 0, 1, and 2. Each injection consists of 5ml solution (10mg/ml). The injection is administered at specific sites in the uterine cavity, including the anterior, posterior, left, right, and fundal walls, or surrounding the suspected lesion area.
  Arms: Experimental Group
Drug: High-dose Progestin — Participants in the control group will receive standard-of-care treatment with oral high-dose progestin alone. The dosage will be Medroxyprogesterone Acetate 250mg-500mg/day or Megestrol Acetate 160mg-320mg/day, taken daily throughout the treatment period
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if intrauterine injection of "Recombinant Humanized Type III Collagen Lyophilized Fibers" works to treat endometrial cancer or atypical hyperplasia in patients seeking fertility-preserving treatment. It will also learn about the safety of this intervention.The main questions it aims to answer are:

1. Does the combination of recombinant humanized type III collagen and progestin significantly increase the tumor remission rate at 6 months compared to progestin alone?
2. What medical problems do participants have when receiving this treatment (e.g., allergic reactions, abnormal inflammatory markers, or histocompatibility issues)? Researchers will compare "recombinant humanized type III collagen plus progestin (experimental group)" to "high-dose progestin alone (control group)" to see if the combination therapy is more effective for fertility preservation.

Participants will:

1. Take high-dose progestin (such as Medroxyprogesterone Acetate or Megestrol Acetate) orally every day.
2. If assigned to the experimental group, receive one intrauterine submucosal injection of collagen via hysteroscopy at months 0, 1, and 2, for a total of 3 injections.
3. Visit the clinic once every 3 months for treatment evaluation and follow-up, which includes hysteroscopic endometrial biopsy, imaging (such as transvaginal ultrasound), and safety tests for relevant biochemical indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of endometrioid adenocarcinoma (G1 or G2) or atypical endometrial hyperplasia.
2. For patients with endometrial cancer, magnetic resonance imaging (MRI) or ultrasound must confirm that the lesion is confined to the endometrium or invades less than 1/2 of the myometrium (i.e., FIGO 2009 Stage IA).
3. Age ≤ 45 years.
4. Desire to preserve fertility and signed informed consent.
5. No serious medical comorbidities (e.g., severe liver or renal dysfunction).
6. No contraindications to progestin therapy or pregnancy.
7. No evidence of distant metastasis on imaging.

Exclusion Criteria:

1. Tumor invasion > 1/2 of the myometrium, or FIGO (2009) Stage IB and above.
2. Tumor differentiation grade G3 or non-endometrioid adenocarcinoma.
3. Coexistence of other malignant tumors.
4. Contraindications to conservative treatment or use of the study drugs.
5. Known allergy to recombinant protein components.
6. Acute genital tract inflammation or untreated abnormal vaginal discharge within 2 weeks prior to enrollment.
7. Previous treatment with high-potency progestin for more than 1 month.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
6-month Tumor Complete Remission Rate | 6 months after the start of treatment

SECONDARY OUTCOMES:
Time to Complete Response (CR) | Up to 2 years
  The duration from the start of treatment to the first documentation of Complete Response (CR), based on negative pathological biopsy and clear imaging findings.
1-Year Recurrence Rate | 1 year after CR
  The proportion of participants who experience disease recurrence within 12 months after achieving Complete Response. Recurrence is defined as reappearance of cancer evidence in pathology or imaging.
Endometrial Thickness and Blood Flow | Every 3 months during the 9-month treatment period
  Evaluation of endometrial thickness (mm) and blood flow status (via Doppler) assessed by transvaginal ultrasound.
1-Year Pregnancy Rate | 1 year after treatment completion
  The percentage of participants who achieve clinical pregnancy within one year following the end of treatment.
Incidence of Adverse Events (Safety) | Throughout the 9-month treatment period
  Monitoring for adverse events, including allergic reactions (rash, itching), systemic inflammatory markers (Complete Blood Count, C-Reactive Protein), and organ function (liver and kidney function tests).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
General clinical data and fertility-sparing treatment outcomes of patients in both the experimental and control groups will be shared.
Supporting Information: Study Protocol
Time Frame: The data will be available within 6 months after the publication of the primary research paper.
Access Criteria: Researchers interested in obtaining the clinical and treatment data can apply by contacting the principal investigator.